CLINICAL TRIAL: NCT03917875
Title: Computer-Delivered Personalized Feedback Intervention for Hazardous Drinkers With Elevated Anxiety Sensitivity
Brief Title: Computer-Delivered PFI for Anxiety Sensitivity/Alcohol Intervention for Hazardous Drinkers With Elevated Anxiety Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, Daniel Paulus, Graduate Student, University of Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00001045
Record Dates: First submitted 2019-04-05; First posted 2019-04-17 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Alcohol Drinking; Anxiety; Coping Behavior
MeSH Terms: conditions — Alcohol Drinking; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- PFI (Experimental)
  Interventions: Behavioral: Personalized feedback intervention

INTERVENTIONS:
Behavioral: Personalized feedback intervention — The novel integrated PFI will be developed and modeled from past PFIs targeting hazardous drinking. Participants will view feedback on the computer screen. The computer program/algorithm will determine the proper normative feedback to participants.
  Arms: PFI

SUMMARY:
Hazardous alcohol consumption is one of the leading causes of preventable deaths in the United States. Further, it is highly comorbid with anxiety and depressive symptoms and disorders; hazardous alcohol use is associated with increased anxiety/depression. Indeed, 'affectively-vulnerable hazardous drinkers' (i.e., drinkers with elevated negative mood states or psychopathology) are 'at risk' for higher drinking rates, more problematic drinking, worsened mental health, and greater disability. Specialty care options are needed to address the unique 'affective needs' of hazardous drinkers. One promising intervention approach is to employ personalized feedback interventions (PFI). These interventions are brief, efficient, and have been shown to be effective in a number of settings and across an array of populations. However, PFIs have not been evaluated among affectively vulnerable hazardous drinkers.

In order to address the heterogeneity of negative mood states and disorders among hazardous drinkers, there is a need to theoretically orient the intervention approach on underlying transdiagnostic processes that underpin affective psychopathology. Anxiety sensitivity (AS), the tendency to fear anxiety-related sensations, is a core transdiagnostic vulnerability factor underlying the etiology and maintenance of anxiety disorders, other emotional disorders, and hazardous drinking. AS is malleable in response to psychosocial interventions, making it a prime risk factor to target in prevention/intervention programs, including PFI approaches. Integrated treatments that address hazardous drinking via AS are nonexistant. As most hazardous drinkers typically do not access treatment because of such barriers as cost, time commitments, stigma, and logistics (e.g., travel, scheduling appointments), there is a need to develop an accessible, brief, integrated tool to explicitly address the drinking-affective vulnerability comorbidity via AS. To address this public health gap, the current proposal seeks to employ a computer-delivered integrated PFI that directly addresses hazardous drinking-AS in a personalized manner. Hazardous drinkers with elevated AS will be randomly assigned to receive one session of PFI or attention information control with follow-up assessments at one week and one month post-intervention. The PFI will focus on targeted feedback about drinking behaviors, AS, and adaptive coping strategies.

ELIGIBILITY:
Inclusion Criteria:

* elevated anxiety sensitivity, hazardous drinking

Exclusion Criteria:

* current mental health/substance treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Motivation for change | 1 month
  The Alcohol Ladder (Clair et al., 2011). The Alcohol Ladder is a reliable and valid (Hogue, Dauber, & Morgenstern, 2010) measure of motivation to change alcohol use. It contains 10 statements that correspond to stages of change: pre-contemplation (e.g., "I enjoy drinking and have decided I'll never change it. I have no interest in changing the way I drink"), contemplation (e.g., "I rarely think about changing the way I drink, and I have no plans to change it"), preparation (e.g., "I definitely plan to change my alcohol use, and I'm almost ready to make some plans about how to change"), action (e.g., "I have changed my drinking, but I still worry about slipping back. So I need to keep working on the changes I've made), and maintenance (e.g., "I have changed my drinking and will never go back to the way I drank before). Participants select the statement that best corresponds to their current stage of motivation regarding changes in their alcohol use.
Drinks per occasion | 1 month
  Drinks per occasion will be assessed as a ratio of the number of drinks consumed in the past 30 days over the number of drinking occasions reported over the past 30 days.
Anxiety Sensitivity | 1 month
  Anxiety Sensitivity sensitivity will be assessed with the Anxiety Sensitivity Index-3 (ASI-3; Taylor et al., 2007). The ASI-3 is an 18-item self-report measure of anxiety sensitivity. Items (e.g., "It scares me when my heart beats rapidly") are rated on a 5-point Likert-type scale from 0 (very little) to 4 (very much). Items are summed to a total score. The ASI-3 shows good convergent and discriminant validity (Taylor et al., 2007).

SECONDARY OUTCOMES:
Drinking to cope | 1 month
  Drinking to cope will be measured with the Drinking motives questionnaire-revised (DMQ-R; Cooper, 1994). The DMQ-R is a 20-item self-report measure of drinking motives. It contains four subscales: social, enhancement, social pressure/conformity, and coping with anxiety/depression. The coping subscale (e.g., "to forget your worries") will serve as the measure of drinking to cope with emotional symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No